CLINICAL TRIAL: NCT03467308
Title: Identification of New Signaling Pathways Targeting Colorectal Cancer in Egyptian Patients
Brief Title: Signaling Pathways Targeting Colorectal Cancer in Egypt
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Alaaeldeen Kamal Thabet, Principal Investigator, Assiut University
Other Study IDs: CRC18
Record Dates: First submitted 2018-02-20; First posted 2018-03-16 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; TIGAR; TRIM59
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Genes, p53; Glutathione

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue samples and normal intestinal tissue samples from the safety margin around the tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal cancer patients: 50 Patients confirmed histopathologically to have early stages of colorectal cancer.
  Interventions: Genetic: Markers in tissue samples: (TIGAR , TRIM59, P53, AKT, GSH)
- Risky group: 20 risky patients (those with ulcerative colitis, chron's disease, familial adenomatous polyposis).
  Interventions: Genetic: Markers in tissue samples: (TIGAR , TRIM59, P53, AKT, GSH)

INTERVENTIONS:
Genetic: Markers in tissue samples: (TIGAR , TRIM59, P53, AKT, GSH) — The followings markers will be investigated in tissue samples:
  1. TIGAR expression using quantitative real-time polymerase chain reaction (q Rt PCR) and immunohistochemistry.
  2. TRIM59 expression using quantitative real-time polymerase chain reaction (q Rt PCR) and immunohistochemistry.
  P53 expression using immunohistochemistry. P53 nuclear localization is essential for its normal function in growth inhibition or induction of apoptosis.
  * Akt expression using western blot.
  * GSH using chemical methods.

SUMMARY:
Colorectal cancer (CRC) is the third most commonly diagnosed cancer and the second leading cause of cancer-related death worldwide. In Egypt, CRC constitutes 4.2% of all cancers with median age is 50 years old.

DETAILED DESCRIPTION:
The TP53-induced glycolysis and apoptosis regulator (TIGAR) is a transcriptional target of p53. TIGAR functions as a fructose-2,6-bisphosphatase, decreasing the flux through the main glycolytic pathway. Consequently, glucose metabolism diverted into the pentose phosphate pathway (PPP). This results in TIGAR-mediated increase in cellular NADPH production, which contributes to the scavenging of ROS by reduced glutathione and thus a lower sensitivity of cells to oxidative stress-associated apoptosis. PPP also produce ribose phosphate for DNA synthesis and repair that play a role in tumor development and cell survival in tumor microenvironment. A high expression level of TIGAR was observed in cancers such as breast cancer, hepatocellular carcinoma, intestinal cancer, and glioblastoma. These studies suggested that TIGAR may act as an oncogene that support cancer progression.

The tripartite motif containing 59 (TRIM) proteins have been implicated in many biological processes including cell differentiation, apoptosis, transcriptional regulation, and signaling pathways.

It is related to several cancers. The oncogenic effect of TRIM59 on tumor proliferation and migration has been studied in various cancers, including gastric cancer, osteosarcoma, lung and CRC. The biological activity of TRIM59 has been observed to be closely associated with the regulation of P53. TRIM59 interacts with P53, leading to P53 ubiquitination and degradation, and consequently promotes tumor growth and migration. TRIM59 functions as an oncogene in CRC progression. It also activates the PI3K/AKT pathway. Increased activity of this pathway is often associated with tumor progression and resistance to cancer therapies. AKT can control TIGAR protein translation by activation of mTOR.

Targeting TRIM59 inhibition will inhibit PI3K-Akt pathway downregulate TIGAR protein translation. This is in turn downregulates GSH levels, increases ROS production, leading to cell death and blocks the cellular proliferation and survival of cancer cells leading to tumor regression. Therefore, TRIM59 protein can serve as a new potential therapeutic target for CRC.

ELIGIBILITY:
Inclusion Criteria:

* All Patients confirmed histopathologically to have early stages of colorectal cancer.
* Risky group patients (including those with ulcerative colitis, chron's disease, familial adenomatous polyposis).

Exclusion Criteria:

* Patients with previous history of CRC treated with chemotherapy or presence of other types of cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * All Patients confirmed histopathologically to have early stages of colorectal cancer admitted to General Surgery Department -Assiut University Hospital for CRC resection.
  * Risky group patients (including those with ulcerative colitis, chron's disease, familial adenomatous polyposis) undergoing diagnostic colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Measure TIGAR in the study groups. | 1 YEAR
  Measure TIGAR expression in colorectal cancer patients and risky group patients.
Measure TRIM59 in the study groups. | 1Year
  Measure TRIM59 expression in colorectal cancer patients and risky group patients.

SECONDARY OUTCOMES:
Targeting new prognostic and therapeutic markers for colorectal cancer. | 1 year
  Finding a relationship between TIGAR and TRIM 59 expression and PI3K/AKT pathway as a major signaling mechanism in tumorigenesis for targeting new prognostic and therapeutic markers for colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Alaaeldeen Kamal, MD (PhD student), Principal Investigator — Assiut University; Ragaa Hamdy Salama, Professor (MD), Study Director — Assiut University; Maha Ali Essam al-Din, lecturer (MD), Study Director — Assiut University; Marwa AbdelHafiz Abdel Hassan, lecturer (MD), Study Director — Assiut University; Ahmed Ali Abdel Motelb, lecturer (MD), Study Director — Assiut University
Locations (1):
- Assiut University- faculty of medicine -Medical biochemistry department, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang J, Wen J, Tian T, Lu Z, Wang Y, Wang Z, Wang X, Yang Y. GLUT-1 overexpression as an unfavorable prognostic biomarker in patients with colorectal cancer. Oncotarget. 2017 Feb 14;8(7):11788-11796. doi: 10.18632/oncotarget.14352. PMID 28052033
- [Background] Cheung EC, Athineos D, Lee P, Ridgway RA, Lambie W, Nixon C, Strathdee D, Blyth K, Sansom OJ, Vousden KH. TIGAR is required for efficient intestinal regeneration and tumorigenesis. Dev Cell. 2013 Jun 10;25(5):463-77. doi: 10.1016/j.devcel.2013.05.001. Epub 2013 May 30. PMID 23726973
- [Background] Won KY, Lim SJ, Kim GY, Kim YW, Han SA, Song JY, Lee DK. Regulatory role of p53 in cancer metabolism via SCO2 and TIGAR in human breast cancer. Hum Pathol. 2012 Feb;43(2):221-8. doi: 10.1016/j.humpath.2011.04.021. Epub 2011 Aug 4. PMID 21820150
- [Background] Zhao M, Fan J, Liu Y, Yu Y, Xu J, Wen Q, Zhang J, Fu S, Wang B, Xiang L, Feng J, Wu J, Yang L. Oncogenic role of the TP53-induced glycolysis and apoptosis regulator in nasopharyngeal carcinoma through NF-kappaB pathway modulation. Int J Oncol. 2016 Feb;48(2):756-64. doi: 10.3892/ijo.2015.3297. Epub 2015 Dec 17. PMID 26691054
- [Background] Zhou Z, Ji Z, Wang Y, Li J, Cao H, Zhu HH, Gao WQ. TRIM59 is up-regulated in gastric tumors, promoting ubiquitination and degradation of p53. Gastroenterology. 2014 Nov;147(5):1043-54. doi: 10.1053/j.gastro.2014.07.021. Epub 2014 Jul 18. PMID 25046164
- [Background] Liang J, Xing D, Li Z, Shen J, Zhao H, Li S. TRIM59 is upregulated and promotes cell proliferation and migration in human osteosarcoma. Mol Med Rep. 2016 Jun;13(6):5200-6. doi: 10.3892/mmr.2016.5183. Epub 2016 Apr 25. PMID 27121462
- [Background] Zhan W, Han T, Zhang C, Xie C, Gan M, Deng K, Fu M, Wang JB. TRIM59 Promotes the Proliferation and Migration of Non-Small Cell Lung Cancer Cells by Upregulating Cell Cycle Related Proteins. PLoS One. 2015 Nov 24;10(11):e0142596. doi: 10.1371/journal.pone.0142596. eCollection 2015. PMID 26599082
- [Background] Sun Y, Ji B, Feng Y, Zhang Y, Ji D, Zhu C, Wang S, Zhang C, Zhang D, Sun Y. TRIM59 facilitates the proliferation of colorectal cancer and promotes metastasis via the PI3K/AKT pathway. Oncol Rep. 2017 Jul;38(1):43-52. doi: 10.3892/or.2017.5654. Epub 2017 May 22. PMID 28534983
- [Background] Ahmad R, Alam M, Hasegawa M, Uchida Y, Al-Obaid O, Kharbanda S, Kufe D. Targeting MUC1-C inhibits the AKT-S6K1-elF4A pathway regulating TIGAR translation in colorectal cancer. Mol Cancer. 2017 Feb 2;16(1):33. doi: 10.1186/s12943-017-0608-9. PMID 28153010